CLINICAL TRIAL: NCT01840839
Title: Impact of Transcranial Slow Oscillating Stimulation on Memory Consolidation During Slow Wave Sleep in Older Adults
Brief Title: Effects of Brain Stimulation During a Daytime Nap on Memory Consolidation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Agnes Flöel, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nap-tSOS-aged
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Older Adults (50-90 Years)
Keywords: aging; cognitive decline; brain stimulation; tSOS; tDCS; sleep; nap; daytime sleep; memory; memory consolidation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0,75 Hz stimulation (Experimental): transcranial slow oscilliating stimulation (tSOS)during periods of SWS
  Interventions: Device: brain stimulation
- no stimulation (Sham Comparator): Sham stimulation during periods of SWS
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: brain stimulation
  Other Names: oscillating direct current brain stimulation
  Arms: 0,75 Hz stimulation
Device: Sham Stimulation
  Other Names: no stimulation
  Arms: no stimulation

SUMMARY:
The beneficial effect of nocturnal as well as daytime sleep on memory consolidation is well-documented in young, healthy subjects. Slow wave sleep (SWS), in particular, with its slow oscillating activity have shown to enhance declarative, hippocampus-dependent memory representations. This impact of sleep on memory performance can be additionally enhanced by exogeneous induction of transcranial slow oscillating stimulation (tSOS) within the frequency range of SWS in humans (0,7- 0,8 Hz) during sleep, as has been demonstrated in young, healthy subjects. If older adults that commonly experiencing cognitive decline, including long-term retention of declarative memory - benefit from transcranial slow oscillatory stimulation (tSOS) during sleep in the same way has not been studied so far. The primary goal of the study is therefore to investigate the impact of oscillating current stimulation (tSOS) during a daytime nap on declarative memory consolidation in older adults.

ELIGIBILITY:
Inclusion Criteria:

* age: 50-90 years
* right handed
* inobtrusive neuropsychological examination

Exclusion Criteria:

* untreated severe internal or psychiatric diseases
* epilepsy
* other severe neurological diseases eg., previous major stroke, brain tumour
* dementia
* contraindications to MRI

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Retention of declarative memories after 0.75 Hz stimulation during SWS, vs after sham stimulation during SWS | 4 weeks
  Retention between stimulation conditions (0.75 Hz during SWS, vs sham stimulation during SWS) in the declarative memory task.

SECONDARY OUTCOMES:
1. Amount of Slow wave Sleep | 4 weeks
  1. Amount of slow wave sleep assessed by standard polysomnographic criteria in 0,75 Hz vs SHAM stimulation during SWS.
2. sleep spindels | 4 weeks
  2.Spindel activity during sleep indicated via several spindel parameters like number, duration, frequency of spindles; compared between 0,75 Hz and SHAM stimulation during SWS.
3. EEG-correlates | 4 weeks
  3. Neuronal correlates (EEG-power in slow oscillation frequency bands induced by 0,75 Hz vs SHAM stimulation during SWS; EEG-correlates of encoding and retrieval of a declarative memory task).
4. further memory systems | 4 weeks
  4. Performance in further memory systems (procedural), compared between 0,75 Hz and SHAM stimulation during SWS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Study Chair — Charite Universitätsmedizin Berlin - Neurologie; Agnes Flöel, Professor, Principal Investigator — Charite Universitätsmedizin Berlin - Neurologie
Locations (1):
- Charite CCM Neurologie Berlin, Berlin, Germany

REFERENCES:
- [Background] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Background] Naismith SL, Lewis SJ, Rogers NL. Sleep-wake changes and cognition in neurodegenerative disease. Prog Brain Res. 2011;190:21-52. doi: 10.1016/B978-0-444-53817-8.00002-5. PMID 21531243
- [Background] Mednick SC, Cai DJ, Kanady J, Drummond SP. Comparing the benefits of caffeine, naps and placebo on verbal, motor and perceptual memory. Behav Brain Res. 2008 Nov 3;193(1):79-86. doi: 10.1016/j.bbr.2008.04.028. Epub 2008 May 8. PMID 18554731
- [Background] Mander BA, Santhanam S, Saletin JM, Walker MP. Wake deterioration and sleep restoration of human learning. Curr Biol. 2011 Mar 8;21(5):R183-4. doi: 10.1016/j.cub.2011.01.019. No abstract available. PMID 21377092
- [Background] Mednick S, Nakayama K, Stickgold R. Sleep-dependent learning: a nap is as good as a night. Nat Neurosci. 2003 Jul;6(7):697-8. doi: 10.1038/nn1078. PMID 12819785
- [Result] Ladenbauer J, Kulzow N, Passmann S, Antonenko D, Grittner U, Tamm S, Floel A. Brain stimulation during an afternoon nap boosts slow oscillatory activity and memory consolidation in older adults. Neuroimage. 2016 Nov 15;142:311-323. doi: 10.1016/j.neuroimage.2016.06.057. Epub 2016 Jul 2. PMID 27381076
- [Derived] Ladenbauer J, Ladenbauer J, Kulzow N, Floel A. Memory-relevant nap sleep physiology in healthy and pathological aging. Sleep. 2021 Jul 9;44(7):zsab002. doi: 10.1093/sleep/zsab002. PMID 33406266